CLINICAL TRIAL: NCT06170918
Title: Half Effective Dose of Remimazolam to Prevent Cardiovascular Response to Tracheal Intubation When Combined With Fentanyl
Brief Title: Dose of Remimazolam in Children for Intubation
Acronym: DRIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XJH-A-20231120
Record Dates: First submitted 2023-11-30; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Anesthesia
Keywords: anesthesia induction; remimazolam; tracheal intubation; median effective dose
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Intervention Model Description: The initial dose is 0.4mg/kg and the dose interval is 0.2mg/kg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- remimazolam (Experimental): Remimazolam is given for anesthesia induction. The initial dosage is 0.4mg/kg, and the interval dosage is 0.02mg/kg.
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — remimazolam is given intravenously
  Other Names: remimazolam besylate

SUMMARY:
Remimazolam has demonstrated the potential as a valuable medication for procedural sedation and general anesthesia. However, half effective dose of remimazolam required to prevent cardiovascular response to tracheal intubation when combined with fentanyl in pediatric patients is still unknown.

ELIGIBILITY:
Inclusion Criteria:

* age from 3 to 12 years old
* patients scheduled for surgery under general anesthesia
* Body mass index in the range of 5% -95% of the same age group
* Consent was obtained from the patient and the family members, and an informed consent form was signed

Exclusion Criteria:

* American Society of Anesthesiologists status ≥3
* patients who cannot cooperate with intravenous anesthesia induction
* patients with risk of difficult airway
* patients who are allergic to benzodiazepines
* patients with neurological dysfunction
* Participate involved in other clinical investigators within 3 months

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
half effective dose for intubation | from injection of remimazolam to completed tracheal intubation, at an average of 5 minutes
  half effective dose of remimazolam required to prevent cardiovascular response to tracheal intubation when combined with fentanyl
cardiovascular response to tracheal intubation | from injection of remimazolam to 3 minutes after tracheal intubation, at an average of 8 minutes
  cardiovascular response is defined as increase of blood pressure or heart rate higher than 20% of the baseline value by 3 minutes after intubation

SECONDARY OUTCOMES:
the time to loss of consciousness | from injection of remimazolam to loss of consciousness, at an average of 3 minutes
incidence of adverse events | from injection of remimazolam to loss of consciousness, at an average of 3 minutes
  adverse events include bradycardia, hypotension, hypoxemia, and injection pain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fang YB, Wang CY, Gao YQ, Cai YH, Chen J, Zhang XL, Dong LQ, Shang-Guan WN, Liu HC. The safety and efficacy of remimazolam tosylate for induction and maintenance of general anesthesia in pediatric patients undergoing elective surgery: Study protocol for a multicenter, randomized, single-blind, positive-controlled clinical trial. Front Pharmacol. 2023 Feb 10;14:1090608. doi: 10.3389/fphar.2023.1090608. eCollection 2023. PMID 36843931
- [Background] Kimoto Y, Hirano T, Kuratani N, Cavanaugh D, Mason KP. Remimazolam as an Adjunct to General Anesthesia in Children: Adverse Events and Outcomes in a Large Cohort of 418 Cases. J Clin Med. 2023 Jun 8;12(12):3930. doi: 10.3390/jcm12123930. PMID 37373624